CLINICAL TRIAL: NCT05566613
Title: Prediction of Individual Radiosensitivity During Radiotherapy for Breast Cancer Patients, the Role of Genetic and Inflammatory Markers
Brief Title: Prediction of Individual Radiosensitivity During Radiotherapy for Breast Cancer Patients
Acronym: SENS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Karolinska University Hospital (Other)
Collaborators: Stockholm University (Other)
Responsible Party: Principal Investigator, Mattias Hedman, Head of Radiotherapy, Karolinska University Hospital
Other Study IDs: 21/079
Record Dates: First submitted 2022-06-12; First posted 2022-10-04 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Radiation Tolerance; Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Single nucleotide polymorphisms (SNPs) will be analysed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Blood sample — Blood sample before and after radiotherapy and photography before radiotherapy

SUMMARY:
Non-randomized clinical cohort study investigating if single nucleotide polymorphism (SNP) or inflammatory markers can predict radiosensitivity in breast cancer patients receiving radiotherapy.

DETAILED DESCRIPTION:
Objectives

1. To explore if acute radiation response can be predicted in patients, by analyzing a single nucleotide polymorphism (SNP rs1801516) sampled prior to radiotherapy.
2. If acute radiation response can be predicted in patients, by analyzing genetic and inflammatory markers in blood sampled prior to radiotherapy.
3. If late side effects from radiotherapy can be predicted in patients, by analyzing genetic and inflammatory markers in blood sampled before and after radiotherapy.
4. If there is a correlation between genetic and inflammatory markers in blood and patient reported outcome measures (PROM) and quality of life (QoL).
5. To train an algorithm to correlate the appearance of skin before radiotherapy and the extent of skin reaction to radiotherapy

Outline This study is a non-randomized clinical cohort study. Adults with breast cancer will be invited to participate in the study. Blood will be collected before start of treatment and after radiotherapy is completed. Quality of life (QoL) and symptoms will be assessed before and weekly during treatment, at the end of treatment and after one year. A total of 550 patients is expected to be recruited.

ELIGIBILITY:
Inclusion criteria:

* Patients receiving adjuvant radiotherapy for breast cancer 2,67 Gy x 15 (or a radio biologically equivalent dose)
* > 18 years
* Being able to read and understand patient information in Swedish
* Signed informed consent

Exclusion criteria:

* Ongoing infection
* Fever >37,9 degrees Celsius
* Unable to follow study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving postoperative radiotherapy for breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2022-05-09 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Acute radiation dermatitis grading criteria | Before and during treatment and after one year
  Acute radiation dermatitis grading criteria according to the Radiation Therapy Oncology Group. Minimum value 1 and maximum value 4, higher value means a worse outcome

SECONDARY OUTCOMES:
Quality of life (QoL) | Before and during treatment and after one year
  Quality of life determined by European Organisation for Research and Treatment of Cancer questionnaire QLQ-C30
Breast cancer specific Quality of life (QoL) | Before and during treatment and after one year
  Quality of life determined by European Organisation for Research and Treatment of Cancer questionnaire QLQ-BR23
Cancer related fatigue Quality of life (QoL) | Before and during treatment and after one year
  Quality of life determined by European Organisation for Research and Treatment of Cancer questionnaire QLQ-FA12
Number of participants with heart disease | at five years
  Heart disease as described in patient chart diagnosed after radiotherapy
Number of participants with lung disease | at five years
  Lung disease as described in patient chart diagnosed after radiotherapy and related to the radiotherapy treatment area

CONTACTS AND LOCATIONS:
Overall Officials: Mattias Hedman, MD PhD, Principal Investigator — Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden